CLINICAL TRIAL: NCT03416569
Title: The Effects of Prazosin on the Attention-Enhancing Effects of Nicotine in Healthy Non-Smokers
Brief Title: Effects of Prazosin on the Attention-Enhancing Effects of Nicotine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unanticipated staff changes are preventing completion within funding period.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Britta Hahn, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00078832
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: no Condition, Basic Science
MeSH Terms: interventions — Nicotine; Prazosin

STUDY DESIGN:
Intervention Model Description: Each participant is tested with each of four test conditions, in counterbalanced sequence.
Masking Description: The study will be double-blind. Only the statistician performing randomization and the dispensing pharmacist will know the sequence of test conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotine-Prazosin Interaction Study (Experimental): Over four test days, each participant will be tested with placebo, nicotine alone, prazosin alone, and nicotine + prazosin, in a double-blind sequence.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Prazosin; Drug: Nicotine + Prazosin

INTERVENTIONS:
Drug: Placebo — placebo skin patch + placebo capsule
Drug: Nicotine — nicotine patch (7 mg/24 hrs) + placebo capsule
Drug: Prazosin — placebo patch (7 mg/24 hrs) + prazosin capsule (1 mg)
Drug: Nicotine + Prazosin — nicotine patch (7 mg/24 hrs) + prazosin capsule (1 mg)

SUMMARY:
To test whether specific aspects of the attention-enhancing effects of nicotine may be mediated by down-stream activation of alpha1 adrenoceptors, the interaction of nicotine and the alpha1 adrenergic antagonist prazosin on cognitive task performance will be tested in human non-smokers. The effects of a low-dose nicotine patch vs. a placebo patch will be tested in the presence and absence of prazosin over 4 test sessions.

DETAILED DESCRIPTION:
Drugs that activate nicotinic acetylcholine receptors (nAChRs), such as nicotine, have cognitive enhancing, and in particular attention-enhancing effects that may be of clinical benefit to individuals with cognitive deficits, such as those diagnosed with Alzheimer's disease, schizophrenia, or ADHD. nAChR agonists can increase the release of other neurotransmitters in the brain, including dopamine, noradrenaline, serotonin, glutamate and GABA. To date, it is unknown which of these actions is central to mediating the attention-enhancing effects of nAChR agonists. Such knowledge would channel drug development efforts onto subtypes of the nAChR expressed on and activating the target system, but not systems such as the subcortical dopamine system involved in unwanted effects of nAChR agonists (e.g., dependence).

Preclinical studies have suggested that the noradrenergic system is critical to the attention-enhancing effects of the prototypical nAChR agonist nicotine. Activation of alpha1-adrenergic receptors appears to be involved in broadening the attentional window, an effect shared with nicotine. The aim of the present study is to test whether the effects of nicotine on broad monitoring may be mediated by alpha1 adrenoceptors by testing the interaction of nicotine and the predominantly alpha1 adrenergic antagonist prazosin in healthy human non-smokers. The effects of a low-dose nicotine patch vs. a placebo patch will be tested in the presence and absence of prazosin in a 2 x 2 within-subject design, over 4 repeated test sessions, in healthy never-smokers. Each participant is asked to complete for test session, on separate days. In each session, a skin patch will be applied and a capsule given by mouth. In one session, both are a placebo. In another session, the patch contains nicotine (7 mg/24 hrs) and the capsule is a placebo. In another session, the patch is a placebo and the capsule contains 1 mg of prazosin. In another session, the patch contains nicotine and the capsule contains prazosin. The sequence of these testing conditions is counterbalanced and double-blind.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 55 years.
* Smoked no more that 40 cigarettes, cigars or cigarillos in lifetime.
* Smoked no cigarettes, cigars or cigarillos in the last year.
* No exposure to any nicotine-containing product in the last month.
* Normal or corrected to normal vision (at least 20/80).

Exclusion Criteria:

* Pregnant or breast-feeding.
* Drug or alcohol abuse or dependence currently or in the last 2 years.
* DSM Axis I mood, anxiety or psychotic disorder.
* Cardiovascular or cerebrovascular disease.
* Hypertension (resting systolic BP above 150 or diastolic above 95 mm Hg).
* Hypotension (resting systolic BP below 90 or diastolic below 60).
* Bradycardia (heart rate <60 bpm).
* Impaired liver or kidney function.
* Severe asthma.
* Obstructive pulmonary disease.
* Type I diabetes.
* Use of any centrally active medications.
* Use of any cardiovascular drugs, including blood pressure medications and antiarrhythmics.
* Use of diuretic medication.
* History of or current neurological illnesses, such as stroke, seizure disorders, neurodegenerative diseases, or organic brain syndrome.
* Learning disability, mental retardation, or any other condition that impedes cognition.
* Planned eye surgery.
* Inability to perform the Rapid Visual Information Processing Task.
* Known hypersensitivity to prazosin, any quinazolines, or nicotine.
* Narcolepsy.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Spatial Attentional Resource Allocation Task reaction time | 5 hrs after patch application (=2.5 hr after ingestion of capsule)
  average reaction time of trials with a signal detection response
Spatial Attentional Resource Allocation Task omission errors | 5 hrs after patch application (=2.5 hr after ingestion of capsule)
  percentage of trials on which no response was registered
Rapid Visual Information Processing Task hit rate | 5 hrs after patch application (=2.5 hr after ingestion of capsule)
  percentage of targets detected
Rapid Visual Information Processing Task reaction time | 5 hrs after patch application (=2.5 hr after ingestion of capsule)
  average reaction time on trials with a correct response
Change Detection Task accuracy | 5 hrs after patch application (=2.5 hr after ingestion of capsule)
  percentage of correct responses
Change Detection reaction time | 5 hrs after patch application (=2.5 hr after ingestion of capsule)
  average reaction time across trials

SECONDARY OUTCOMES:
Blood pressure | hourly for 8 hours on each test day
  mmHg
Vital signs: heart rate | hourly for 8 hours on each test day
  beats per minute

IPD SHARING:
Plan to Share IPD: No